CLINICAL TRIAL: NCT05341531
Title: Relationship Between Perioperative Related Factors and Inflammatory Markers and Postoperative Delirium in Elderly Patients With Non-cardiac Major Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bijia Song, principal investigator, Beijing Friendship Hospital
Other Study IDs: Risk factors and delirium
Record Dates: First submitted 2022-03-17; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Preoperative Sleep Disorder; Preoperative Anxiety; Inflammatory Reaction; Postoperative Delirium
MeSH Terms: conditions — Inflammation; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: elderly patients undergoing non-cardiac surgery — Elderly patients 60 years and older undergoing major non-cardiac surgery > 2 hours

SUMMARY:
Perioperative neurocognitive impairment, including postoperative delirium (POD), is common in older patients after anesthesia and surgery and is associated with poorer short- and long-term outcomes, including worsening cognitive decline, surgical Complications, increased risk of hospitalization, and death after cardiac and noncardiac surgery. POD is more common with age, occurs in up to 65% of elderly patients, and increases in patients with mild cognitive impairment. As more and more older adults undergo surgery and anesthesia, POD has become a major global health challenge requiring urgent attention. Prevention strategies involving multidisciplinary perioperative interventions may have some benefit overall, but the impact on POD remains uncertain. Known inflammatory responses may be associated with adverse outcomes such as neurocognitive dysfunction and cancer recurrence after major surgery. Different anesthesia methods, the regulation of anesthesia drugs on postoperative inflammatory response has been confirmed in vitro, but its clinical significance is still unclear. Therefore, exploring the risk factors of inducing POD has important clinical significance for the early prevention of POD. Second, a recent study found that the incidence of POD was significantly higher in patients whose sleep cycle was disturbed during hospitalization. Animal experiments found that after 5 hours of sleep deprivation in adult mice, the number of dendritic spines in CA1 neurons in the hippocampus was reduced, and the length of dendrites was significantly shortened, which damaged the synaptic transmission of the central nervous system, and significantly improved memory and cognitive function. Damaged. And many studies have investigated whether bispectral index (BIS)-guided anesthesia is associated with a reduced risk of POD, compared with "standard-of-care" anesthesia or the use of goal-directed end-tidal volatile agent concentrations, the reasoning is that the use of BIS-guided anesthesia results in less anesthesia exposure, and therefore "light" anesthesia may reduce the incidence of postoperative POD compared to "deep" anesthesia. However, this conclusion is still controversial. The study of Anshentong et al. has confirmed that deep anesthesia with BIS maintained at 40-49 can delay postoperative recovery time, reduce the level of inflammatory factors and the incidence of early postoperative cognitive impairment, and reduce the incidence of early postoperative cognitive impairment. Brain damage. Therefore, although age is known to be the main correlative factor for POD, different depths of anesthesia may cause different stress responses in patients, resulting in different release of inflammatory factors. An additional risk factor may be preoperative psychiatric symptoms, and assessment of mental status is often overshadowed by concerns about multiple comorbidities in older adults. Anxiety disorders are one of the prominent psychiatric symptoms in older adults. very common. Preoperative anxiety is defined as an unpleasant restless or tense state secondary to patient concerns about illness, hospitalization, anesthesia, surgery, or the unknown. Studies on the relationship between preoperative anxiety and POD also vary in consistency due to the characteristics of different populations. Many of the current studies are mostly single-center with limited sample size, which may have a certain bias in the conclusions. Therefore, the investigators designed and planned to conduct a multi-center, large-sample cohort study to determine the impact of perioperative related factors and inflammatory markers on elderly patients undergoing non-cardiac major surgery .

ELIGIBILITY:
Inclusion Criteria:

* ①patients over 60 years old;

  * ASA grade II-IV;

    * major surgery for >2 hours,

      * hospital stay >2 days.

Exclusion Criteria:

* ①History of neurological, cerebral or psychiatric diseases;

  * History of alcoholism or drug dependence;

    * Preoperative delirium, or previous postoperative delirium; ④No obvious visual, auditory, and communication impairment;

      * No obvious liver and kidney Functional impairment; ⑥ The surgical site interferes with BIS electrode placement;

        * Planned wake-up test during the surgery; ⑧ No follow-up is expected after 1 year.

Ages: 60 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elderly patients 60 years and older undergoing major non-cardiac surgery > 2 hours
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative cognitive function | one day before surgery
  The Mini Mental Scale (MMSE) assessed cognitive function at baseline. The evaluation items of MMSE include: location, attention, computing ability of asking time and place, immediate recall ability of short-term review language, and graph reproduction ability. The test is conducted in the way of asking questions. The scale score ranges from 0 to 30 points, and the final score is 27-30 points, which can be regarded as normal. If the score is less than 27 points, it can be regarded as cognitive impairment.
Perioperative cognitive function | first day after surgery
  The Confusion Assessment Method (CAM) assessed cognitive function on the first day after surgery.
Perioperative cognitive function | third day after surgery
  The Confusion Assessment Method (CAM) assessed cognitive function on the third day after surgery.
Perioperative cognitive function | one week after surgery
  The Confusion Assessment Method (CAM) assessed cognitive function on the day of discharge
Perioperative cognitive function | 30 days after surgery
  Minimal Telephone Scale (AMTS) assessed cognitive function at 30 days after surgery, and 1 year after surgery, respectively. Scores 6 or below have been shown to correlate well with dementia.
Perioperative cognitive function | 1 year after surgery
  Minimal Telephone Scale (AMTS) assessed cognitive function at 30 days after surgery, and 1 year after surgery, respectively. Scores 6 or below have been shown to correlate well with dementia.
preoperative sleep quality | 24 hours before surgery
  The Pittsburgh Sleep Quality Index (PSQI) scale was used to evaluate the patient's sleep status 24 hours before surgery for sleep quality during the past month.The Pittsburgh sleep quality index was assessed by 19 self-rated questions and 5 sleep peers problem composition. Only 19 self-rated questions were scored. The 19 self-assessment questions consist of 7 of 03 points. A factor. "0" means no difficulty and "3" means very difficult. All factors are added to form 021. Total score of the scale. "0" means no difficulty and "21" means very difficulty in all aspects
postoperative sleep quality | first day after surgery
  Postoperative sleep scores were recorded using the Athens Insomnia Scale (AIS). 0-3 means no insomnia 4-6 means suspected insomnia. >6 insomnia
postoperative sleep quality | third day after surgery
  Postoperative sleep scores were recorded using the Athens Insomnia Scale (AIS). 0-3 means no insomnia 4-6 means suspected insomnia. >6 insomnia
preoperative anxiety | one day before surgery
  The preoperative anxiety level was assessed by the Hans Anxiety Scale (HADS) before the operation. 0-3 means no insomnia 4-6 means suspected insomnia. >6 insomnia

SECONDARY OUTCOMES:
patients characteristics | one day before surgery
  Record the patient's characteristics before surgery
surgery characteristics | during the surgery
  Record the patient's surgery characteristics during operation
perioperative inflammatory markers: systemic inflammation index (SII) | baseline before surgery
  SII=platelet count×neutrophil count/lymphocyte count
perioperative inflammatory markers: systemic inflammation index (SII) | first day after surgery
  SII=platelet count×neutrophil count/lymphocyte count
perioperative inflammatory markers: systemic inflammation index (SII) | third day after surgery
  SII=platelet count×neutrophil count/lymphocyte count
perioperative inflammatory markers: neutrophil-to-lymphocyte ratio (NLR) | baseline before surgery
  NLR=neutrophil count/lymphocyte count
perioperative inflammatory markers: neutrophil-to-lymphocyte ratio (NLR) | first day after surgery
  NLR=neutrophil count/lymphocyte count
perioperative inflammatory markers: neutrophil-to-lymphocyte ratio (NLR) | third day after surgery
  NLR=neutrophil count/lymphocyte count
perioperative inflammatory markers: monocyte-to-lymphocyte ratio (MLR) | baseline before surgery
  MLR=monocyte count/lymphocyte count
perioperative inflammatory markers: monocyte-to-lymphocyte ratio (MLR) | first day after surgery
  MLR=monocyte count/lymphocyte count
perioperative inflammatory markers: monocyte-to-lymphocyte ratio (MLR) | third day after surgery
  MLR=monocyte count/lymphocyte count
perioperative inflammatory markers: c-reactive protein ( CRP) | baseline before surgery
  markers: c-reactive protein ( CRP)
perioperative inflammatory markers: c-reactive protein ( CRP) | first day after surgery
  markers: c-reactive protein ( CRP)
perioperative inflammatory markers: c-reactive protein ( CRP) | third day after surgery
  markers: c-reactive protein ( CRP)